CLINICAL TRIAL: NCT04785222
Title: The Effects of Infraorbital Nerve Block With Dexmedetomidine Added to Bupivacaine on Fentanyl Requirement During Endoscopic Transsphenoidal Approach to Remove Pituitary Tumor: Prospective Randomized Double Blinded Control Study
Brief Title: Infraorbital Nerve Block for Endoscopic Transsphenoidal Approach to Remove Pituitary Tumor
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Pathomporn Pin on, M.D., Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ANE_04032021
Record Dates: First submitted 2021-03-03; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Intraoperative Pain Control
Keywords: Infraorbital nerve block; Endoscopic Transsphenoid Approach; Pituitary tumors
MeSH Terms: conditions — Pituitary Neoplasms | interventions — Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: Intervention and group assignment: The subjects will be randomized into three groups, as following.
  Group DB: Bilateral infraorbital nerve block with dexmedetomidine 5 mcg mixed with 0.5% plain bupivacaine, in total volume of 2 ml per side Group BP: Bilateral infraorbital nerve block with 0.5% plain bupivacaine, a volume of 2 ml per side Group NS (control): Bilateral infraorbital nerve block with normal saline 2 ml per side
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The outside of the envelope is an individual code (e.g., IC2, CY1). Inside an envelope is a group (DB, BP, or NS). A nurse will prepare local anesthetics in a two 3-ml syringe and put them in the envelope according to the allocation order. The syringe will be containing the same volume of clear drugs which are unable to be distinguished between groups.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- DB (Experimental): Group DB: Bilateral infraorbital nerve block with dexmedetomidine 5 mcg mixed with 0.5% plain bupivacaine, in total volume of 2 ml per side
  Interventions: Drug: dexmedetomidine 5 mcg mixed with 0.5% plain bupivacaine
- BP (Active Comparator): Group BP: Bilateral infraorbital nerve block with 0.5% plain bupivacaine, a volume of 2 ml per side
  Interventions: Drug: dexmedetomidine 5 mcg mixed with 0.5% plain bupivacaine
- NS (Placebo Comparator): Group NS (control): Bilateral infraorbital nerve block with normal saline 2 ml per side
  Interventions: Drug: dexmedetomidine 5 mcg mixed with 0.5% plain bupivacaine

INTERVENTIONS:
Drug: dexmedetomidine 5 mcg mixed with 0.5% plain bupivacaine — Bilateral infraorbital nerve block with dexmedetomidine 5 mcg mixed with 0.5% plain bupivacaine, in total volume of 2 ml per side
  Other Names: DB

SUMMARY:
Perioperative pain relief during endoscopic transsphenoidal pituitary surgery is generally treated with opioids either morphine sulfate or fentanyl. This study will compare the traditional method of intravenous fentanyl to the bilateral infraorbital nerve block in adult patients scheduled for pituitary surgery by the transsphenoidal approach.

DETAILED DESCRIPTION:
1. Infraorbital nerve- The infraorbital nerve exits from the infraorbital foramen. It is a branch of the maxillary nerve, the second division of the trigeminal nerve, the fifth cranial nerve. The infraorbital nerve is a pure sensory nerve innervates the lateral aspect of the nose, upper lip, upper incisor, canines, premolars, and the first molar of the ipsilateral side. (1-6) The NYSORA website mentions that 'transsphenoidal hypophysectomy' is one of the indications of infraorbital nerve block. (2) There are two approaches to block this nerve, the intraoral and extraoral approaches. Regardless to the approach, the infraorbital foramen must be palpated throughout the procedure to avoid the serious complication of eyeball penetration. (2,4,6) This study, we use the extraoral approach with a 27-gauge needle advance perpendicularly toward the foramen. When the bony resistance is appreciated, slowly injects 2 ml of local anesthetics. After the injection, gently massage over the puncture site to prevent the hematoma formation. (2)
2. Pituitary adenomas- Pituitary adenomas are the tumors of the pituitary gland. The tumors can be classified by the size and/ or by the functional status of hormone production. Dimension < 1 cm is microadenoma and dimension ≥ 1 cm is called macroadenoma. (7) Treatment options for pituitary tumors are surgery, radiation, and medications. The single or combination of treatment depends on types of tumor, its size, how fast the tumor grows, patient's age, and patient's general condition. (8) The two main surgical techniques for removing pituitary tumors are endoscopic trans-nasal transsphenoidal (ETSS) approach and transcranial or craniotomy approach. The transsphenoidal approach has many advantages such as less brain tissue damage than those in craniotomy approach. There is no visible scar because a small incision will be done over the nasal septum and through the sphenoid sinus. The bony posterior wall of sphenoid sinus is drilled with small surgical chisels to reach the pituitary gland. (9) Choice of anesthesia for ETSS approach is general anesthesia with cuffed endotracheal intubation strap over the left corner of patient's mouth. Balanced anesthetic technique is maintained throughout the surgical procedure. Specific goals for ETSS pituitary surgery are optimized hormonal function, facilitate surgical exposure, surveillance and promptly treatment for massive bleeding from accidentally penetration to the cavernous sinus. General goals for neurosurgery are maintain the hemodynamic stability and rapid emergence. (10) Promoting selective nerve block instead of systemic opioid analgesics, we anticipate to see a rapid wear off from general anesthesia and rapid awakening.
3. Characteristics of pain in pituitary adenomas - A cross-sectional study of 278 patients with pituitary adenomas was shown that i) the prevalence of somatic pain (called 'bodily pain' in the study) was high and independent to the tumor type, ii) the patients diagnosed of Cushing's disease were more susceptible to pain than the patients diagnosed of other pituitary diseases, iii) a high incidence of headache which is independent to the tumor type, and iv) pain significantly correlated to depression and quality of life (QoL).(11,12) Pituitary tumor headache was reported unilaterally, at the site of orbital and retro-orbital, and throbbing in quality. Its severity was moderate to strong. (12) According to International Headache Society (IHS), pituitary tumor caused chronic and episodic migraine, 46% and 30%, respectively. (13,14) These findings demonstrate the importance of adequate pain relieve during pituitary surgery while rapid awakening after general anesthesia is required.
4. Dexmedetomidine addition to bupivacaine - Addition of dexmedetomidine to bupivacaine in greater palatine nerve block and supra-zygomatic maxillary nerve block was resulted prolong the analgesic duration, decrease postoperative analgesic requirement, and no additional side effects such as hemodynamic disturbance and sedation. (15,16) The reported dosage was 0.5-1 µg/kg of dexmedetomidine. A systematic review of nine RCTs revealed many positive effects of dexmedetomidine in facilitating neuraxial and peripheral nerve block. (16) Dexmedetomidine-related adverse effects were transient bradycardia in brachial plexus block but did not observe in intrathecal administration. Respiratory depression was not seen. A high dosage of dexmedetomidine (15 µg) administered intrathecally caused higher sedation level during surgery. (17) The result from this study will add more evidence of the use of perineural dexmedetomidine in clinical setting.

Materials and methods Study hypothesis: We hypothesize that the bilateral infraorbital nerve block with dexmedetomidine added to bupivacaine reduce fentanyl used during endoscopic transsphenoidal pituitary surgery.

Study design: Prospective randomized double blinded control (patients and assessors will be blinded) Participants: Adult patients, age ≥ 18 years old, diagnosis of pituitary tumor, scheduled for endoscopic transsphenoidal approach to remove tumor under general anesthesia with endotracheal tube.

The exclusion criteria will be 1) the patient is known case of allergy to dexmedetomidine, 2) the patient allergy to bupivacaine, 3) the patient does not sign a consent form to participate to the study, 4) the operation is changed due to cavernous sinus perforation, 5) the navigator and Mayfield is used to identify the tumor There are no pre-specified withdrawal criteria. The expected duration of subject participation is 3 days including the surgical day, which is day-1. At the time of pre-surgical evaluation and informed consent, participants will be informed that their participation in this research is voluntary and they may discontinue participation without consequence at any time. The data obtained prior to the subject's decision of withdrawal will be retained and analyzed in consistent with the study purpose. Unless the participants indicate that they want to remove their data from the study.

Ethical consideration: Before commencement of the study, the research proposal must be approved by the Ethical Committee (EC) of Faculty of Medicine, Chiang Mai University (CMU). The protocol will be registered to the Research Operation System (ROS) and the website www.clinicaltrial.gov. Participants of this study should be fully level of conscious, E4V5M6. The research team will explain the procedure and risks to the participants one day prior to the surgery. If the participants decide to be enrolled, the consent form will be asked to sign.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* age ≥ 18 years old
* diagnosis of pituitary tumor
* scheduled for endoscopic transsphenoidal approach to remove tumor under general anesthesia with endotracheal tube

Exclusion Criteria:

* the patient is known case of allergy to dexmedetomidine
* the patient allergy to bupivacaine
* the patient does not sign a consent form to participate to the study
* the operation is changed due to cavernous sinus perforation
* the navigator and Mayfield is used to identify the tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The total fentanyl used (mcg) during the endoscopic transsphenoidal pituitary surgery. | in operating room during surgery
  fentanyl administered iv during surgery according to the criteria of vital sign changes

SECONDARY OUTCOMES:
Time to the second dose of i.v. fentanyl | during surgery
  after the first dose of fentanyl given in all patients, the duration for the second dose according to the vital sign changes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mariano ER, Watson D, Loland VJ, Chu LF, Cheng GS, Mehta SH, Maldonado RC, Ilfeld BM. Bilateral infraorbital nerve blocks decrease postoperative pain but do not reduce time to discharge following outpatient nasal surgery. Can J Anaesth. 2009 Aug;56(8):584-9. doi: 10.1007/s12630-009-9119-5. Epub 2009 May 28. PMID 19475468
- [Background] Kaushal A, Haldar R. Regional Anesthesia in Neuroanesthesia Practice. Discoveries (Craiova). 2020 Jun 29;8(2):e111. doi: 10.15190/d.2020.8. PMID 32637571
- [Background] Ezzat S, Asa SL, Couldwell WT, Barr CE, Dodge WE, Vance ML, McCutcheon IE. The prevalence of pituitary adenomas: a systematic review. Cancer. 2004 Aug 1;101(3):613-9. doi: 10.1002/cncr.20412. PMID 15274075
- [Background] Dunn LK, Nemergut EC. Anesthesia for transsphenoidal pituitary surgery. Curr Opin Anaesthesiol. 2013 Oct;26(5):549-54. doi: 10.1097/01.aco.0000432521.01339.ab. PMID 23963232
- [Background] Dimopoulou C, Athanasoulia AP, Hanisch E, Held S, Sprenger T, Toelle TR, Roemmler-Zehrer J, Schopohl J, Stalla GK, Sievers C. Clinical characteristics of pain in patients with pituitary adenomas. Eur J Endocrinol. 2014 Nov;171(5):581-91. doi: 10.1530/EJE-14-0375. Epub 2014 Aug 12. PMID 25117460